CLINICAL TRIAL: NCT06406608
Title: Patient-derived Organoid Drug Sensitivity Guided Treatment for Drug-resistant Recurrent Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Kingbio Medical (Beijing) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-107
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organoid-Guided therapy (Experimental): All patients will be included in a single-arm. Participants will undergo biopsy of tumor tissue for subsequent organoid generation and drug sensitivity tests.
  Interventions: Other: Chemotherapy and targeted-therapy guided by organoid drug sensitivity test

INTERVENTIONS:
Other: Chemotherapy and targeted-therapy guided by organoid drug sensitivity test — This study conducts drug sensitivity tests on various clinically approved drugs. The most sensitive drug for the patient is selected for treatment. This study aims to evaluate the clinical effectiveness of treatment plans guided by organoid drug sensitivity tests.

SUMMARY:
This study aims to enroll non-small cell lung cancer patients who have undergone at least two rounds of standard treatment for drug resistance/recurrence. Patient-derived Organoid will be established, and drug sensitivity test will be conducted to intervene in the selection of clinical treatment plans. Efficacy evaluation and prognosis analysis will also be conducted. It is hoped that this study will provide a basis for the development of personalized treatment plans.

DETAILED DESCRIPTION:
Twenty patients with drug-resistant/relapsed non-small cell lung cancer who met the inclusion criteria were enrolled in the study after signing an informed consent form. Tumor samples were obtained through clinical puncture, and qualified samples were subjected to organoid modeling. Perform drug sensitivity test on the established lung cancer organoids. The drugs used are all that have been marketed and applied in clinical practice. According to the results of organoid drug sensitivity analysis, the patient received a treatment plan with relatively sensitive drugs. Follow up prognostic data and relevant clinical information of enrolled patients, conduct statistical analysis on the consistency between drug sensitivity test results and patient treatment response, and evaluate the clinical effectiveness of treatment plans guided by organoid drug sensitivity results.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years old (calculated based on the date of signing informed consent);
2. Diagnosed as drug-resistant/relapsed non-small cell lung cancer;
3. After at least two systemic treatments and the disease progresses;
4. According to the efficacy evaluation criteria of solid tumors (RECIST 1.1), at least one lesion that has not received radiation therapy, has not received other local therapies, and can obtain tumor tissue (can be from a single lesion source or multiple lesions combined) is used for organoid establishment;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1;
6. Expected survival time>3 months;
7. Before a tumor sample can be taken, there must be a record of disease progression on imaging after the previous treatment.;
8. The patient has informed consent and signed a written consent form;
9. The patients had good compliance and willingly followed the study plan, including scheduled visits, treatments, laboratory tests, and other research steps.

Exclusion Criteria:

1. Extremely weakened overall condition, unable to tolerate bronchoscopy examination;
2. Patients with acute suppurative inflammation of the respiratory tract accompanied by high fever, acute asthma attacks, and ongoing hemoptysis;
3. Have a history of interstitial lung disease, non infectious pneumonia or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc
4. Patients with active leptomeningeal disease or brain metastasis;
5. Diagnosed with other malignant diseases other than NSCLC within 5 years prior to initial administration (excluding curative basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or curative resection of carcinoma in situ);
6. Have a history of immunodeficiency, including positive HIV serum tests;
7. Active hepatitis B without treatment (defined as HBsAg positive and HBV-DNA copy number detected is greater than the upper limit of normal value in the laboratory of the research center);
8. The presence of any serious or uncontrollable systemic diseases;
9. Pregnant or lactating female patients;
10. The researchers believe that patients who are not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1-2 years
  Percentage of patient's measurable disease who have achieved either complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Progressive free survival | 1-2 years
  The time from initiation of treatment to the occurrence of disease progression or death.
Overall survival time | 2 years
  The time from the date of randomization to the date of death for any cause. Patients will be followed until their date of death or until final database closure.

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, PhD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Background] Carney DN. Lung cancer--time to move on from chemotherapy. N Engl J Med. 2002 Jan 10;346(2):126-8. doi: 10.1056/NEJM200201103460211. No abstract available. PMID 11784881
- [Background] Kashima J, Kitadai R, Okuma Y. Molecular and Morphological Profiling of Lung Cancer: A Foundation for "Next-Generation" Pathologists and Oncologists. Cancers (Basel). 2019 Apr 29;11(5):599. doi: 10.3390/cancers11050599. PMID 31035693
- [Background] Zhang Z, Yang S, Ma Y, Zhou H, Wu X, Han J, Hou J, Hao L, Spicer JD, Koh YW, Provencio M, Reguart N, Mitsudomi T, Wang Q. Consistency of recommendations for the diagnosis and treatment of non-small cell lung cancer: a systematic review. Transl Lung Cancer Res. 2021 Jun;10(6):2715-2732. doi: 10.21037/tlcr-21-423. PMID 34295672
- [Background] Muto S, Inomata S, Yamaguchi H, Mine H, Takagi H, Watanabe M, Ozaki Y, Inoue T, Yamaura T, Fukuhara M, Okabe N, Matsumura Y, Hasegawa T, Osugi J, Hoshino M, Higuchi M, Shio Y, Suzuki H. [Resistance Mechanisms to Immune Checkpoint Inhibitor and Its Overcome with Focus on beta-Catenin in Lung Cancer]. Gan To Kagaku Ryoho. 2022 Sep;49(9):928-931. Japanese. PMID 36156007
- [Background] Seidlitz T, Merker SR, Rothe A, Zakrzewski F, von Neubeck C, Grutzmann K, Sommer U, Schweitzer C, Scholch S, Uhlemann H, Gaebler AM, Werner K, Krause M, Baretton GB, Welsch T, Koo BK, Aust DE, Klink B, Weitz J, Stange DE. Human gastric cancer modelling using organoids. Gut. 2019 Feb;68(2):207-217. doi: 10.1136/gutjnl-2017-314549. Epub 2018 Apr 27. PMID 29703791
- [Background] Romero-Calvo I, Weber CR, Ray M, Brown M, Kirby K, Nandi RK, Long TM, Sparrow SM, Ugolkov A, Qiang W, Zhang Y, Brunetti T, Kindler H, Segal JP, Rzhetsky A, Mazar AP, Buschmann MM, Weichselbaum R, Roggin K, White KP. Human Organoids Share Structural and Genetic Features with Primary Pancreatic Adenocarcinoma Tumors. Mol Cancer Res. 2019 Jan;17(1):70-83. doi: 10.1158/1541-7786.MCR-18-0531. Epub 2018 Aug 31. PMID 30171177
- [Background] Li M, Izpisua Belmonte JC. Organoids - Preclinical Models of Human Disease. N Engl J Med. 2019 Feb 7;380(6):569-579. doi: 10.1056/NEJMra1806175. No abstract available. PMID 30726695
- [Background] Kim SY, Kim SM, Lim S, Lee JY, Choi SJ, Yang SD, Yun MR, Kim CG, Gu SR, Park C, Park AY, Lim SM, Heo SG, Kim H, Cho BC. Modeling Clinical Responses to Targeted Therapies by Patient-Derived Organoids of Advanced Lung Adenocarcinoma. Clin Cancer Res. 2021 Aug 1;27(15):4397-4409. doi: 10.1158/1078-0432.CCR-20-5026. Epub 2021 Jun 3. PMID 34083237
- [Background] Wang HM, Zhang CY, Peng KC, Chen ZX, Su JW, Li YF, Li WF, Gao QY, Zhang SL, Chen YQ, Zhou Q, Xu C, Xu CR, Wang Z, Su J, Yan HH, Zhang XC, Chen HJ, Wu YL, Yang JJ. Using patient-derived organoids to predict locally advanced or metastatic lung cancer tumor response: A real-world study. Cell Rep Med. 2023 Feb 21;4(2):100911. doi: 10.1016/j.xcrm.2022.100911. Epub 2023 Jan 18. PMID 36657446
- [Background] Drost J, Clevers H. Organoids in cancer research. Nat Rev Cancer. 2018 Jul;18(7):407-418. doi: 10.1038/s41568-018-0007-6. PMID 29692415